CLINICAL TRIAL: NCT05324956
Title: The Relationship Between Bone Mineral Density With Respiratory Functions and Exercise Capacity in Postmenopausal Women
Brief Title: The Relationship Between Bone Mineral Density With Respiratory Functions and Exercise Capacity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Öykünur CANSU, Principal investigator, Izmir Bakircay University
Other Study IDs: 2021/348
Record Dates: First submitted 2022-02-22; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Postmenopausal Women
Keywords: Osteopenia; Osteoporosis; Spirometry; 6 Minute Walk Test; New York Posture Rating Chart
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postmenopausal Women: Postmenopausal women be between 40-79 years and being diagnosed with osteoporosis or osteopenia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Individuals will not receive any interventions

SUMMARY:
If the bone mineral density of a patient with a diagnosis of osteopenia falls further, he develops osteoporosis.Menopause causes many changes in women's bodies in the form of vasomotor, sleep disorders, fatigue, aches and pains, altered cognitive functions, as well as genitourinary problems such as vaginal dryness, irritation, recurrent urinary tract infections. In the long term, inevitable changes occur in the musculoskeletal system. Osteoporosis, sarcopenia, postural dysfunction, regression in gait cycle, Loss of balance control and instability and increased risk of falling are the changes reported during this period. These mentioned effects negatively affect the quality of life of women. The aim of this study is to investigate the relationship of bone mineral density with respiratory functions and exercise capacity in postmenopausal women.The second aim is to compare the respiratory functions and exercise capacities of postmenopausal women with osteopenia and osteoporosis.

DETAILED DESCRIPTION:
The 1993 Consensus Development Conference paper defined osteoporosis as ''a disease characterized by low bone mass and microarchitectural deterioration of bone tissue, leading to increased bone fragility and consequent increased risk of fracture.In 1994, the World Health Organization (WHO) established criteria for measuring bone mineral density (BMD) that allowed the diagnosis of osteoporosis before fractures. This practical definition is based on the main (known) risk factor: reduced bone strength or density and people at high risk but without fractures.Premenopausal women have a low rate of osteoporosis; however, the prevalence increases with age due to progressive bone loss.Bone densitometry is an established method for evaluating osteoporosis. Various different methods have been developed in the last 25 years. DEXA is recommended and FDA approved for BMD measurement; It is precise, noninvasive, has low radiation exposure and takes 10 minutes to administer. Osteoporosis can have a significant impact on patients' daily lives. Vertebral deformity causes loss of spinal mobility, and patients with osteoporosis have difficulty standing, bending over, getting up from a chair, walking, carrying objects, dressing, fixing hair, bathing, moving in bed, using the toilet, and descending to the floor. Compared with women without existing vertebral deformities, women with extensive deformities have higher crude mortality and hospitalization rates overall.Osteoporosis deprives older women of many of their social roles. Failure to fulfill roles such as cooking, housework, work, and intimacy can be devastating, leading to frustration and embarrassment. Interpersonal relationships can be deeply affected by the effects of osteoporosis, straining family ties and destroying extra-familial relationships, leading to social isolation. Therefore, treatment options should be well evaluated because affected individuals should focus not only on bone remodeling, but also on ways in which negative outcomes such as pain, depression and loss of self-esteem can be improved. Considering all these situations, we asked the question whether there is any relationship between bone mineral density and respiratory functions and exercise capacity. In order to evaluate these parameters, we decided to examine the patient's detailed demographic information, posture evaluation according to the New York Posture Scale, 6-minute walking test result, and Pulmonary Function Test result.

ELIGIBILITY:
Inclusion Criteria:

* Between 40-80 years old
* Female gender
* Being diagnosed with menopause
* Being diagnosed with osteoporosis or osteopenia
* Volunteer to participate in the study

Exclusion Criteria:

* Hemoptysis of unknown cause
* Recent abdominal, thoracic, or eye surgery
* Thoracic, abdominal, or cerebral aneurysm
* pulmonary embolism
* Mental state disorder that interferes with cooperation
* Arrhythmias disrupting hemodynamics
* Having any diagnosed disease affecting the respiratory system
* pneumothorax
* unstable angina
* Recent myocardial infarction
* Thrombosis in lower extremity
* Acute myocarditis
* Other diseases that will prevent exercise (infection, kidney failure)

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women aged between 40-80 years old and diagnosed with osteoporosis or osteopenia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Respiratory Functions | at baseline
  Spirometry will be applied to evaluate respiratory functions.It is the most commonly performed lung function test, which evaluates volume against time using a device called a spirometer. The expiratory time should be at least 6 seconds and extended up to 15 seconds if necessary.The patient is instructed to take a deep breath and blow as hard and as fast as possible and take a deep breath to complete the flow volume cycle. The one with the highest values out of at least three tests done in succession is selected.
Evaluation of Exercise Capacity | at baseline
  6 Minutes Walking Test will be applied to evaluate exercise capacity. The goal of this test is to walk the maximum distance that can be walked in 6 minutes. Average walking distances: 20/50 age:590-640m 60/70 age:540/570m 70/80 age:470-530m.
Posture Assessment | at baseline
  Posture assessment will be made using the New York Posture Rating Chart (NYPR).NYPR is an inexpensive, easy and fast-applied subjective postural assessment method that is widely used for clinical postural assessment. The grading chart is used to evaluate 13 areas of the body based on the assumption that posture is the alignment of the body and its parts.Each field is awarded a point based on position: 5 points for correct position; 3 points for a slight deviation and 1 point for a significant deviation. The total score ranges from 18-90 points. The higher the score, the better the postural alignment.

CONTACTS AND LOCATIONS:
Locations (1):
- Öykünur CANSU, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided